CLINICAL TRIAL: NCT05427123
Title: A Collaborative Treatment Network for Youth With or at High Risk for Bipolar Disorder
Brief Title: Children's Bipolar Network Treatment Trial I
Acronym: CBN
Status: Recruiting | Type: Observational
Sponsor: University of California, Los Angeles (Other)
Collaborators: University of Pittsburgh (Other); Virginia Commonwealth University (Other); University of Colorado, Denver (Other); Milken Institute (Other); Baszucki Brain Research Fund (Other)
Responsible Party: Principal Investigator, David J. Miklowitz, Ph.D., Distinguished Professor of Psychiatry, University of California, Los Angeles
Other Study IDs: IRB#22-000309
Record Dates: First submitted 2022-03-18; First posted 2022-06-22 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Bipolar Disorder; Bipolar I Disorder; Bipolar II Disorder; Other Specified Bipolar and Related Disorder; Mood Instability; Child Mental Disorder; Adolescent - Emotional Problem
Keywords: medication; psychosocial; treatment; longitudinal; naturalistic; assessment
MeSH Terms: conditions — Bipolar Disorder; Neurodevelopmental Disorders | interventions — Dosage Forms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Specimens (i.e., blood samples) obtained for routine lab testing (assays of C-Reactive Protein) will be discarded or destroyed once used for the purposes described in the protocol.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Youth with or at clinical high risk for Bipolar Spectrum Disorder: Youth included in the study will have a Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (DSM-5) diagnosis of Bipolar I or II, Cyclothymic Disorder, or Other Specified Bipolar Disorder (per Course and Outcome of Bipolar Youth study definition)
  Interventions: Other: Medication or psychosocial treatment

INTERVENTIONS:
Other: Medication or psychosocial treatment — Youth included in this naturalistic study will be offered medication management from study psychiatrists. The study's Network Oversight Committee, consisting of PI psychiatrists and consultants, has created guidelines on best practice medications, dosing, and adjustments for the study. The Network Oversight Committee will also offer ongoing consultation to study psychiatrists. The treating physician will take these guidelines and recommendations under consideration but will use clinical judgment and have the final say, in consultation with the parents and child, as to what treatments are prescribed. While psychosocial interventions are of interest as a predictor of outcomes, no universal psychotherapy or other psychosocial treatment will be provided by sites. There is no limitation on participant enrollment in psychosocial treatments. Investigators and their clinical partners may offer these interventions based on clinical judgment and availability.

SUMMARY:
This is a naturalistic treatment and follow-up study of youth with bipolar spectrum disorders (BSDs) across four US sites of The Childhood Bipolar Network (CBN). CBN sites have expertise in diagnosing, assessing, and treating BSDs in youth. The primary aims of this study are to (1) identify and reliably diagnose youth (ages 9 to 19 yrs) with full bipolar disorder (BD) and BSDs, and (2) examine predictors (e.g., mood instability, inflammatory marker C-reactive protein) of clinical outcome over a 12 month period. Participating youth will initially complete a screening that includes a structured diagnostic interview and a baseline blood draw to measure inflammatory processes. Youth with BSD and parents (80 families) will be asked to participate in multiple follow up research visits with interviews, rating instruments, and questionnaires. Per established CBN guidelines, study psychiatrists will provide and track medication management and sites will also track psychosocial treatments. This study ultimately aims to further understanding of best practice pediatric BSD psychiatric and psychosocial treatments and development of a standardized and validated set of clinical tools for patient assessment, diagnosis, and tracking.

DETAILED DESCRIPTION:
Study Background and Significance

Cross-site research networks for specific childhood diseases have led to important treatment advances, such as guidance of optimizing treatments for individual patients and significant reductions in childhood mortality. The Childhood Bipolar Network (CBN) is a similar type of research collaboration developed to support advancements to the understanding and treatment of pediatric bipolar spectrum disorders (BSDs), starting with this first study. The study builds on recent advances in the early identification and reliable diagnosis of pediatric BSDs. It also builds on advances in treatment for youth with or at high risk for BSD, such as the finding from randomized clinical trials showing that family intervention plus pharmacotherapy is consistently associated with superior symptomatic, suicidal, and functional outcomes compared with either usual care or supportive therapy plus pharmacotherapy.

Specific Aims of the Study

The aims of the first study with 80 youth are to (1) identify and reliably diagnose diverse youth (9 to 19 yrs) with BSD I, II, and Other Specified Bipolar Disorder (OSBD, formerly called Bipolar Disorder Not Otherwise Specified) across collaborative clinics in the US; and (2) examine predictors of 1-year treatment response in youth with BSDs, using treatment methods and instrumentation harmonized across four sites. This study will examine mood instability and an inflammatory marker based on a blood test (C-reactive protein) as primary predictors of outcomes.

Study phases and outcomes include: I. Recruitment and screening, II. Intake (blood draw, medical history, structured diagnostic interview, youth mood symptom and instability measures, youth and family functioning measures), III. Weekly parent online reporting on youth symptoms and functioning, IV. Follow-up at 6 and 12 months for repeated measures and relevant updates.

Study milestones will include cross-site harmonization of assessment and treatment methods, validation of a mood instability phenotype, and development of an open trial infrastructure for novel treatments for youth with or at risk for BSD. The development of a standardized BSD clinical assessment and care procedure across US centers is critical to the broader effort to develop robust treatment algorithms and empirically based guidelines for use in a wide variety of national and international health care settings with culturally heterogeneous populations of youth with or at risk for BSD.

ELIGIBILITY:
Inclusion Criteria:

* Youth 9-19 years old
* Youth diagnosed with Bipolar disorder (I, II, Other Specified) or Cyclothymic Disorder by the study team during the diagnostic interview screening
* Youth is able to read and communicate in English to the degree necessary to be able to assent and participate (with help) in their treatment and assessments appropriate for ages 9 and up
* Youth has a caregiver able to participate in ongoing basis in assessment and treatment
* The participating caregiver can reliably read and communicate in English for purposes of study consenting, assessment, and treatment, unless preferred language translation services are regularly available.

Exclusion Criteria:

* Youth has DSM-5 diagnosis of autism spectrum disorder
* Youth has DSM-5 diagnosis of substance or alcohol abuse with impairment within 3 mos.
* Youth has a medical or psychiatric disorder that is life-threatening or requires immediate hospitalization or emergency medical or therapeutic treatment
* Evidence of recent sexual or physical abuse of the youth by legally responsible caregivers
* Evidence of recent intimate partner violence between caregivers responsible for the youth's care

Ages: 9 Years to 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Participants will be recruited and followed through the University of California, Los Angeles (UCLA) Child and Adolescent Mood Disorders Program. Some families elected to be contacted directly about future studies such as this one during general screening or consenting for prior studies. Participants will also be recruited under similar protocols at additional study sites including the Virginia Treatment Center for Children (VTCC) and University of Pittsburgh Child and Adolescent Bipolar Spectrum Services (CABS). Participants at University of Colorado Anschutz Medical Campus study site will be recruited from the Johnson Depression Center and Summit Child Clinic.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2022-07-01 (Actual); Primary Completion 2027-01-01 (Estimated); Study Completion 2027-07-01 (Estimated)

PRIMARY OUTCOMES:
Change in Adolescent Longitudinal Interval Follow-up Evaluation (A-LIFE) Psychiatric Status Ratings | The measure will be administered at 0, 6, and 12 months.
  The A-LIFE is a measure of severity of youth mood symptoms and episodes, including first episode onset, duration, recovery, and recurrence. Independent evaluators administer the A-LIFE interview to the youth and one parent, and rate each week of the prior 6 month interval (i.e., 6 months prior to intake) on Psychiatric Status Ratings (PSRs) of depression, hypomania, mania, and suicidality. The minimum and maximum Psychiatric Status Ratings values are 0 and 6 respectively, with higher Psychiatric Status Ratings meaning worse psychiatric severity.
Change in Children's Affective Lability Scale (CALS), Child and Parent Report forms | The measure will be administered at 0, 6, and 12 months.
  CALS is a measure of youth mood lability and yields subscores for elevation/activation, irritability, and anxiety-depression. It consists of 20 items covering the prior 3 months: "Suddenly becomes tense or anxious…has bursts of being overly affectionate or silly….starts to laugh or cry…suddenly appears sad, depressed, for no reason." The CALS uses a five level Likert scale, from 0 (never or rarely occurs) to 4 (occurs 1 or more times a day). Total score for the 20 items can vary from 0 to 80, with lower scores indicating a lesser degree of affective lability.
Change in Conflict Behavior Questionnaire (CBQ) scores, Child and Parent Report forms | The measure will be administered at 0, 6, and 12 months.
  The CBQ assesses the degree of aversive communication and conflict experienced in a child/parent dyad over the prior 3 months. The 20 scale items are rated "true/false" and cover argumentativeness (e.g., "At least three times a week, we get angry at each other"), frustration in communication, degree of empathy (e.g., "My mother understands me"), and relationship quality (e.g. "I don't think we get along very well"). The child fills out separate CBQs regarding conflict with each primary caregiver. Total scores range from 0 to 20. Higher scores represent more conflict including negative communications.
Kiddo-KINDL Quality of Life Questionnaire for Children, Child and Parent Reports forms | The measure will be administered at 0, 6, and 12 months.
  This Kiddo-KINDL is a measure of youth quality of life in five domains (Emotional Well-being, Self-esteem, Family, Social Contacts, School). Items (e.g., "I did things together with my friends") are rated by the adolescent and parent on a Likert scale from 1 (never) to 5 (all the time) for the past week. The parent form contains items that pertain to the youth's quality of life while the child form pertains to the youth patient. Subscales represent each domain with scores range from 4 to 20. Total scale scores range from 20 to 100. Higher scores on subscales or the total scale mean greater quality of life.

SECONDARY OUTCOMES:
Change in Parents' Online Weekly Evaluation and Rating Scale (POWERS), Parent Report form | The measure will be administered at 0 months and then weekly through 12 months.
  The POWERS is a measure of the severity of youth psychopathology across several symptom domains. Parents rate six symptom domains (anxiety, depression, attention deficit hyperactivity disorder, oppositional defiance, manic, overall symptoms) on symptom severity (0=none to 3=severe) and frequency (0= rarely to 3= almost all of the time) for the past week. Total scale score ranges from 0 to 36, while symptom severity and frequency subscales each range from 0 to 18. Higher scores represent greater psychopathology.
Change in General Behavior Inventory, Parent Version Short form (P-GBI) | The measure will be administered at 0, 6, and 12 months.
  The P-GBI Mania scale is a measure of youth hypomanic/biphasic symptom severity. An example item is "Has your child's mood or energy shifted rapidly back and forth from happy to sad or high to low?" 10 items are each rated by parents on a Likert scale ranging from 1 (never or hardly ever) to 4 (very often or almost constantly) for the past six months. Total scores range from 10 to 40, with higher scores representing greater youth hypomanic/biphasic symptom severity.
Change in Mood and Feelings Questionnaire (MFQ), Child and Parent Report forms | The measure will be administered at 0, 6, and 12 months.
  The MFQ is a measure of severity of youth suicidal ideation and depression. Example items include "I didn't enjoy anything at all," "I thought about death or dying," and "I slept a lot more than usual." The youth or parent rates 33 items as "not true" (0), "sometimes true (1) or "true" (2) for the past two weeks. Total scores range from 0 to 66, with higher scores representing greater severity of suicidal ideation and depression.
Change in Self-Report for Childhood Anxiety Related Disorders (SCARED), Child Report form | The measure will be administered at 0, 6, and 12 months.
  The SCARED is a measure of severity of youth anxiety severity and types of anxiety or worry. An example item is "When I feel frightened, it is hard to breathe." The 41-items are rated by as "Not True or Hardly Ever True" (0), "Somewhat True or Sometimes True" (1), or "Very True or Often True" (2). Total scores range from 0 to 82, with higher scores representing greater severity of anxiety and worry. A total score of ≥ 25 may indicate the presence of an Anxiety Disorder
Drug Use Screening Inventory, Revised (DUSI-R), Child Report form | The measure will be administered at 0, 6, and 12 months.
  DUSI-R is a measure of frequency and severity of drug and alcohol use for the prior month. Participants are instructed to "darken the circle that applies to the number of times you have used each of the drugs listed below in the last month." Item ratings range from 0=no times to 4=More than 20 times. The youth rates 15 additional severity items as yes (0) or no (1), with an example item being "Have you had a craving or very strong desire for alcohol or drugs?" The interviewer may assist with form completion to ensure understanding and completion. Total severity scale scores range from 0 to 15, with higher scores representing more severe substance use.
Change in Positive and Negative Affect Schedule for Children (PANAS-C-SF), Child Report Short form | The measure will be administered at 0, 6, and 12 months.
  PANAS-C-SF is a measure of youth positive and negative affect. Instructions are to "Please indicate how much you have felt this way over the past 15 minutes," with youth asked to rate eight emotions on 5-point Likert scales from 1=Not much at all to 5=a lot for six consecutive days. Four items comprise the positive affect subscale (joyful, happy, lively, proud) while another four items comprise the negative affect subscale (miserable, mad, scared, sad). Subscale scores range from 4 to 20, with higher scores representing more affect.
Change in Perceived Criticism on Perceived Criticism Scale (PC), Child Report form | The measure will be administered at 0, 6, and 12 months.
  The Perceived Criticism (PC) scale measures severity of perceived parental criticism. Youth make a weekly rating for any primary parental figures of "How critical is your parent of you?" and "When this parent criticizes you, how upset do you get?" on scales ranging from 1 (not at all) to 10 (extremely). Total scores range from 2 to 20 with higher scores representing greater perceived criticism.

CONTACTS AND LOCATIONS:
Overall Officials: David J Miklowitz, PhD, Principal Investigator — University of California, Los Angeles
Locations (4):
- United States (4):
  - University of California, Los Angeles, Max Gray Child and Adolescent Mood Disorders Program (CHAMP), Los Angeles, California
  - University of Colorado Anschutz Medical Campus, Helen and Arthur E. Johnson Depression Center, Aurora, Colorado
  - University of Pittsburgh Child and Adolescent Bipolar Spectrum Services Clinic (CABS), Pittsburgh, Pennsylvania
  - Virginia Commonwealth University Medical Center, Richmond, Virginia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Birmaher B, Khetarpal S, Brent D, Cully M, Balach L, Kaufman J, Neer SM. The Screen for Child Anxiety Related Emotional Disorders (SCARED): scale construction and psychometric characteristics. J Am Acad Child Adolesc Psychiatry. 1997 Apr;36(4):545-53. doi: 10.1097/00004583-199704000-00018. PMID 9100430
- [Background] Birmaher B, Merranko JA, Goldstein TR, Gill MK, Goldstein BI, Hower H, Yen S, Hafeman D, Strober M, Diler RS, Axelson D, Ryan ND, Keller MB. A Risk Calculator to Predict the Individual Risk of Conversion From Subthreshold Bipolar Symptoms to Bipolar Disorder I or II in Youth. J Am Acad Child Adolesc Psychiatry. 2018 Oct;57(10):755-763.e4. doi: 10.1016/j.jaac.2018.05.023. Epub 2018 Aug 7. PMID 30274650
- [Background] Chang KD. Course and impact of bipolar disorder in young patients. J Clin Psychiatry. 2010 Feb;71(2):e05. doi: 10.4088/JCP.8125tx7c. PMID 20193644
- [Background] Costello EJ, Angold A. Scales to assess child and adolescent depression: checklists, screens, and nets. J Am Acad Child Adolesc Psychiatry. 1988 Nov;27(6):726-37. doi: 10.1097/00004583-198811000-00011. No abstract available. PMID 3058677
- [Background] Gerson AC, Gerring JP, Freund L, Joshi PT, Capozzoli J, Brady K, Denckla MB. The Children's Affective Lability Scale: a psychometric evaluation of reliability. Psychiatry Res. 1996 Dec 20;65(3):189-98. doi: 10.1016/s0165-1781(96)02851-x. PMID 9029668
- [Background] Goldstein BI, Birmaher B, Carlson GA, DelBello MP, Findling RL, Fristad M, Kowatch RA, Miklowitz DJ, Nery FG, Perez-Algorta G, Van Meter A, Zeni CP, Correll CU, Kim HW, Wozniak J, Chang KD, Hillegers M, Youngstrom EA. The International Society for Bipolar Disorders Task Force report on pediatric bipolar disorder: Knowledge to date and directions for future research. Bipolar Disord. 2017 Nov;19(7):524-543. doi: 10.1111/bdi.12556. Epub 2017 Sep 25. PMID 28944987
- [Background] Goldstein TR, Birmaher B, Axelson D, Ryan ND, Strober MA, Gill MK, Valeri S, Chiappetta L, Leonard H, Hunt J, Bridge JA, Brent DA, Keller M. History of suicide attempts in pediatric bipolar disorder: factors associated with increased risk. Bipolar Disord. 2005 Dec;7(6):525-35. doi: 10.1111/j.1399-5618.2005.00263.x. PMID 16403178
- [Background] Ebesutani C, Okamura K, Higa-McMillan C, Chorpita BF. A psychometric analysis of the Positive and Negative Affect Schedule for Children-Parent Version in a school sample. Psychol Assess. 2011 Jun;23(2):406-16. doi: 10.1037/a0022057. PMID 21381834
- [Background] Hafeman DM, Merranko J, Goldstein TR, Axelson D, Goldstein BI, Monk K, Hickey MB, Sakolsky D, Diler R, Iyengar S, Brent DA, Kupfer DJ, Kattan MW, Birmaher B. Assessment of a Person-Level Risk Calculator to Predict New-Onset Bipolar Spectrum Disorder in Youth at Familial Risk. JAMA Psychiatry. 2017 Aug 1;74(8):841-847. doi: 10.1001/jamapsychiatry.2017.1763. PMID 28678992
- [Background] Kaufman J, Birmaher B, Brent DA, Ryan ND, Rao U. K-SADS-PL. J Am Acad Child Adolesc Psychiatry. 2000 Oct;39(10):1208. doi: 10.1097/00004583-200010000-00002. No abstract available. PMID 11026169
- [Background] Keller MB, Lavori PW, Friedman B, Nielsen E, Endicott J, McDonald-Scott P, Andreasen NC. The Longitudinal Interval Follow-up Evaluation. A comprehensive method for assessing outcome in prospective longitudinal studies. Arch Gen Psychiatry. 1987 Jun;44(6):540-8. doi: 10.1001/archpsyc.1987.01800180050009. PMID 3579500
- [Background] Kowatch RA, Fristad M, Birmaher B, Wagner KD, Findling RL, Hellander M; Child Psychiatric Workgroup on Bipolar Disorder. Treatment guidelines for children and adolescents with bipolar disorder. J Am Acad Child Adolesc Psychiatry. 2005 Mar;44(3):213-35. doi: 10.1097/00004583-200503000-00006. PMID 15725966
- [Background] Hooley JM, Miklowitz DJ. Perceived Criticism in the Treatment of a High-Risk Adolescent. J Clin Psychol. 2017 May;73(5):570-578. doi: 10.1002/jclp.22454. Epub 2017 Jan 23. PMID 28112810
- [Background] Miklowitz DJ, Efthimiou O, Furukawa TA, Scott J, McLaren R, Geddes JR, Cipriani A. Adjunctive Psychotherapy for Bipolar Disorder: A Systematic Review and Component Network Meta-analysis. JAMA Psychiatry. 2021 Feb 1;78(2):141-150. doi: 10.1001/jamapsychiatry.2020.2993. PMID 33052390
- [Background] Miklowitz DJ, Merranko JA, Weintraub MJ, Walshaw PD, Singh MK, Chang KD, Schneck CD. Effects of family-focused therapy on suicidal ideation and behavior in youth at high risk for bipolar disorder. J Affect Disord. 2020 Oct 1;275:14-22. doi: 10.1016/j.jad.2020.06.015. Epub 2020 Jun 26. PMID 32658817
- [Background] Miklowitz DJ, Schneck CD, George EL, Taylor DO, Sugar CA, Birmaher B, Kowatch RA, DelBello MP, Axelson DA. Pharmacotherapy and family-focused treatment for adolescents with bipolar I and II disorders: a 2-year randomized trial. Am J Psychiatry. 2014 Jun;171(6):658-67. doi: 10.1176/appi.ajp.2014.13081130. PMID 24626789
- [Background] Miklowitz DJ, Schneck CD, Walshaw PD, Singh MK, Sullivan AE, Suddath RL, Forgey Borlik M, Sugar CA, Chang KD. Effects of Family-Focused Therapy vs Enhanced Usual Care for Symptomatic Youths at High Risk for Bipolar Disorder: A Randomized Clinical Trial. JAMA Psychiatry. 2020 May 1;77(5):455-463. doi: 10.1001/jamapsychiatry.2019.4520. PMID 31940011
- [Background] Oh DL, Jerman P, Purewal Boparai SK, Koita K, Briner S, Bucci M, Harris NB. Review of Tools for Measuring Exposure to Adversity in Children and Adolescents. J Pediatr Health Care. 2018 Nov-Dec;32(6):564-583. doi: 10.1016/j.pedhc.2018.04.021. Epub 2018 Jun 29. PMID 30369409
- [Background] Perlick DA, Miklowitz DJ, Link BG, Struening E, Kaczynski R, Gonzalez J, Manning LN, Wolff N, Rosenheck RA. Perceived stigma and depression among caregivers of patients with bipolar disorder. Br J Psychiatry. 2007 Jun;190:535-6. doi: 10.1192/bjp.bp.105.020826. PMID 17541117
- [Background] Post RM, Goldstein BI, Birmaher B, Findling RL, Frey BN, DelBello MP, Miklowitz DJ. Toward prevention of bipolar disorder in at-risk children: Potential strategies ahead of the data. J Affect Disord. 2020 Jul 1;272:508-520. doi: 10.1016/j.jad.2020.03.025. Epub 2020 Mar 6. PMID 32553395
- [Background] Post RM, Rowe M, Kaplan D, Findling R. The Child Network for Parents to Track Their Child's Mood and Behavior. J Child Adolesc Psychopharmacol. 2017 Nov;27(9):840-843. doi: 10.1089/cap.2017.0002. Epub 2017 Apr 25. PMID 28441041
- [Background] Prinz RJ, Foster S, Kent RN, O'Leary KD. Multivariate assessment of conflict in distressed and nondistressed mother-adolescent dyads. J Appl Behav Anal. 1979 Winter;12(4):691-700. doi: 10.1901/jaba.1979.12-691. PMID 541311
- [Background] Ravens-Sieberer U, Bullinger M. Assessing health-related quality of life in chronically ill children with the German KINDL: first psychometric and content analytical results. Qual Life Res. 1998 Jul;7(5):399-407. doi: 10.1023/a:1008853819715. PMID 9691720
- [Background] Scheffer RE, Kowatch RA, Carmody T, Rush AJ. Randomized, placebo-controlled trial of mixed amphetamine salts for symptoms of comorbid ADHD in pediatric bipolar disorder after mood stabilization with divalproex sodium. Am J Psychiatry. 2005 Jan;162(1):58-64. doi: 10.1176/appi.ajp.162.1.58. PMID 15625202
- [Background] Schneck CD, Chang KD, Singh MK, DelBello MP, Miklowitz DJ. A Pharmacologic Algorithm for Youth Who Are at High Risk for Bipolar Disorder. J Child Adolesc Psychopharmacol. 2017 Nov;27(9):796-805. doi: 10.1089/cap.2017.0035. Epub 2017 Jul 21. PMID 28731778
- [Background] Shaffer D, Gould MS, Brasic J, Ambrosini P, Fisher P, Bird H, Aluwahlia S. A children's global assessment scale (CGAS). Arch Gen Psychiatry. 1983 Nov;40(11):1228-31. doi: 10.1001/archpsyc.1983.01790100074010. PMID 6639293
- [Background] Spearing MK, Post RM, Leverich GS, Brandt D, Nolen W. Modification of the Clinical Global Impressions (CGI) Scale for use in bipolar illness (BP): the CGI-BP. Psychiatry Res. 1997 Dec 5;73(3):159-71. doi: 10.1016/s0165-1781(97)00123-6. PMID 9481807
- [Background] Tarter RE. Evaluation and treatment of adolescent substance abuse: a decision tree method. Am J Drug Alcohol Abuse. 1990;16(1-2):1-46. doi: 10.3109/00952999009001570. PMID 2330931
- [Background] Weissman MM, Wickramaratne P, Adams P, Wolk S, Verdeli H, Olfson M. Brief screening for family psychiatric history: the family history screen. Arch Gen Psychiatry. 2000 Jul;57(7):675-82. doi: 10.1001/archpsyc.57.7.675. PMID 10891038
- [Background] Yatham LN, Kennedy SH, Parikh SV, Schaffer A, Bond DJ, Frey BN, Sharma V, Goldstein BI, Rej S, Beaulieu S, Alda M, MacQueen G, Milev RV, Ravindran A, O'Donovan C, McIntosh D, Lam RW, Vazquez G, Kapczinski F, McIntyre RS, Kozicky J, Kanba S, Lafer B, Suppes T, Calabrese JR, Vieta E, Malhi G, Post RM, Berk M. Canadian Network for Mood and Anxiety Treatments (CANMAT) and International Society for Bipolar Disorders (ISBD) 2018 guidelines for the management of patients with bipolar disorder. Bipolar Disord. 2018 Mar;20(2):97-170. doi: 10.1111/bdi.12609. Epub 2018 Mar 14. PMID 29536616
- [Background] Youngstrom EA, Frazier TW, Demeter C, Calabrese JR, Findling RL. Developing a 10-item mania scale from the Parent General Behavior Inventory for children and adolescents. J Clin Psychiatry. 2008 May;69(5):831-9. doi: 10.4088/jcp.v69n0517. PMID 18452343
- See also: UCLA Max Gray Child and Adolescent Mood Disorders Program (CHAMP) Website in Los Angeles, CA — https://www.semel.ucla.edu/champ
- See also: Child and Adolescent Bipolar Spectrum Services (CABS) at Western Psychiatric Institute and Clinic of University of Pittsburgh Medical Center (UPMC) in Pittsburgh, PA — https://www.pediatricbipolar.pitt.edu/
- See also: Virginia Commonwealth University (VCU) Medical Center Cameron K. Gallagher Mental Health Resource Center Virginia Treatment Center for Children (VTCC) — https://www.chrichmond.org/services/mental-health/virginia-treatment-center-for-children

DOCUMENTS (3):
  • Study Protocol (2022-03-01): https://cdn.clinicaltrials.gov/large-docs/23/NCT05427123/Prot_000.pdf
  • Informed Consent Form: Youth (13-19y) and Parent Consent (2022-03-10): https://cdn.clinicaltrials.gov/large-docs/23/NCT05427123/ICF_001.pdf
  • Informed Consent Form: Child (9-12y) Assent (2022-03-10): https://cdn.clinicaltrials.gov/large-docs/23/NCT05427123/ICF_002.pdf